CLINICAL TRIAL: NCT00855569
Title: Use of a HemostaticTextile (StasilonTM) to Control Bleeding at Skin Graft Donor Sites (Randomized, Single-Blind)
Brief Title: Hemostatic Textile to Control Bleeding at Donor Graft Sites
Acronym: Stasilon
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: PREN-101
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2012-06

CONDITIONS: Wounds
Keywords: allografting
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Each donor site will act as it own control - both dressings will be applied to the donor site and assessments will be made
  Interventions: Device: Stasilon

INTERVENTIONS:
Device: Stasilon — Stasilon and gauze will be applied to donor site. Dressings will be collected and evaluated for amount of shed blood.

SUMMARY:
The rationale underlying the study is that donor site bleeding is common and often problematic when presenting to the burn surgeon or staff. Frequently, gauze wound dressings are not sufficiently hemostatic to control a donor site bleed thereby leading to administration of vasoconstrictive agents and repeated application of wound dressing/pressure. The hemostatic textile Stasilon™ has proven superior to gauze in reducing bleeding from anesthetized pigs undergoing standardized surgically-induced trauma. Also, observational case reports have noted cessation of bleeding in a limited number of human patients with difficult to control bleeds.

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years old
* burn injury requiring allografting from donor site

Exclusion Criteria:

* < 18 years
* unable to give consent due to mental or emotional instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the UNC Jaycee Burn Center
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of a new hemostatic textile named Stasilon™ against standard wound dressings in controlling burn patient donor graft site bleeding. | At the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Preston Rich, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Jaycee Burn Center, Chapel Hill, North Carolina, United States